CLINICAL TRIAL: NCT02780206
Title: Omics Profiling of the Response to Food and Variability of Weight Loss in Medically Supervised Very Low Calorie Diet
Brief Title: Very Low Calorie Diet Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2016-0304
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Very Low Calorie Diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- obese (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed. Subjects may sign a medical release form to obtain medical and psychological information about them that will help determine study eligibility or can be used for later coding.
  3 study days (one baseline, one approx 2 weeks of diet, one post-diet): muscle mass and function tests, resting energy expenditure, stable isotope infusions with blood draws, and questionnaires regarding quality of life, mood and depression, diet.
  Interventions: Other: Stable isotope amino acid infusion

INTERVENTIONS:
Other: Stable isotope amino acid infusion — such as glycerol, D2O, tyrosine, phenylalanine, glucose, arginine, and citrulline

SUMMARY:
Understanding how foods and nutrients are digested, absorbed and metabolized when weight is stable and during weight loss induced by very low calorie diet procedure using the technologies of genomics, transcriptomics, proteomics, metabolomics and fluxomics ("omics") will enable generation of new hypotheses that could explain the inter-individual differences in weight loss and could lead to optimization and individualization of therapies designed to lose weight.

DETAILED DESCRIPTION:
The overarching hypothesis is that there are baseline, pre- and post-diet combinations of 'omics' signatures in response to food and nutrients that explain the weight loss response of obese subjects to the very low calorie (VLC) diet.

In order to address the general hypothesis the following specific aims will be addressed:

Specific Aim 1: To test the hypothesis that there is a combination of 'omics' parameters in response to a defined meal that discriminate between morbidly obese subjects.

Specific Aim 2: To test the hypothesis that variation in % weight loss to the 2-weeks of VLC diet is related to baseline genomic markers, gene expression profile, proteomic and metabolomic signatures as well as baseline metabolic and substrates fluxomics response to a defined meal.

Specific Aim 3: To test the hypothesis that variation in % weight loss to the 4-weeks of VLC diet is related to baseline genomic markers, gene expression profile, proteomic and metabolomic signatures as well as baseline metabolic and substrates fluxomics response to a defined meal.

ELIGIBILITY:
Inclusion criteria obese subjects:

Diagnosed with morbid obesity (defined as BMI > 40 kg/m2 or BMI > 35 kg/m2 with at least one serious comorbidity (2013 NIH compendium guidelines)) Scheduled for medically supervised Very Low Calorie Diet Age 30 years and older Ability to lay in supine or elevated position for 5 hours Willingness and ability to comply with the protocol Exclusion Criteria Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy control group only) Participation in Weight Loss Management Program within the last 6 months prior the first study day Presence of fever within the last 3 days Untreated metabolic diseases including hepatic or renal disorder unrelated to the primary disease Presence of acute illness or metabolically unstable chronic illness unrelated to the primary disease

· (Possible) pregnancy Any other condition according to the PI or nurse that would interfere with the study or safety of the patient Failure to give informed consent Use of protein or amino acid containing nutritional supplements within 3 days of first test day

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in net whole-body protein synthesis | 0, 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 225, 240, 260, 280, 300, 320, 340, 360 ± 5 min
  Change in whole-body protein synthesis rate after intake of meal

SECONDARY OUTCOMES:
Group differences in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  a fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Executive Function-Adolescent/Adult Sensory Profile (ASP) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  a standardized self-questionnaire that generates an individualized profile of sensory processing across four quadrants: low registration, sensation seeking, sensory sensitivity, and sensation avoiding.
Group differences in quality of life as measured by Short Form (36) Health Survey (SF36) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  self administered questionnaire that measures each of the following eight health concepts: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); Mental Health (MH) as well as a reported Health Transition item (HT)
Group differences in activity as measured by Physical Activity Scale for the Elderly (PASE) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  questionnaire is intended for use in an elderly population and focuses on 3 types of activities: leisure time activities, household activities and work-related activities.
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  a word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Group differences in state of mood as measured by the Profile of Mood State (POMS) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  A psychological distress scale to measure mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment. Healthy populations take 3 to 7 minutes to complete, and others may take up a bit longer.
Group differences in learning and memory as measured by Controlled Oral Word Association Test (COWAT) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  Controlled Oral Word Association Test (COWAT): The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonetic verbal fluency. The raw score (total and mean words recorded across the three trials) was reported.
Group differences in learning and memory as measured by Auditory Verbal Learning Test (AVLT) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  Auditory Verbal Learning Test (AVLT): a verbal episodic memory test that evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, retention and recognition of information
Group differences in attention and executive functions as measured by PASAT | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability.
Group differences in attention and executive functions as measured by Trail Making Test (TMT) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Group differences in attention and executive functions as measured by Brief-A | Postabsorptive state during 3 hours and change after feeding on study day 1 and the change from day 2 and day 3
  a standardized self-report that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
Skeletal muscle strength | on study day 1 and the change from day 2 and day 3
  handgrip and kin-com 1-leg test
24 hour diet recall | on study day 1 and the change from day 2 and day 3
  The subject is asked to recall in detail all the food and drink consumed during the 24 hours prior to the test day.
Respiratory muscle strength | on study day 1 and the change from day 2 and day 3
  Maximum inhalation and exhalation pressure
Body Composition | on study day 1 and the change from day 2 and day 3
  Body composition as measured by Dual-Energy X-ray Absorptiometry on study day 1 and the change from day 2 and day 3
Gut function | postabsorptive and prandial state every 20 minutes up to 6 hours before each sip feeding on day 1 and the change from day 2 and day 3
  Digestion of the stable tracers of amino acid

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wierzchowska-McNew RA, Engelen MPKJ, Thaden JJ, Ten Have GAM, Deutz NEP. Obesity- and sex-related metabolism of arginine and nitric oxide in adults. Am J Clin Nutr. 2022 Dec 19;116(6):1610-1620. doi: 10.1093/ajcn/nqac277. PMID 36166849